CLINICAL TRIAL: NCT01874964
Title: A Randomized Trail of Continues Methadone Maintenance Versus Detoxification in Jail
Brief Title: Trial of Methadone Maintenance Versus Methadone Detox in Jail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIDA-R01DA027211
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2010-12

CONDITIONS: Opioid-Related Disorders
Keywords: HIV Prevention; Opioid-Related Disorders; Medication Assisted Treatment; Methadone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methadone Maintenance (Experimental): Participants assigned to Arm 1 will be maintained on ther pre-incarceration methadone dosage during short term incarceration (6 months or less) and will be actively transferred back to their community methadone clinic upon release from incarceration. Additionally, the study will pay for the cost of methadone maintenance treatment for 10 weeks after re-enrollment post release.
  Interventions: Behavioral: Methadone Maintenance
- Methadone Detoxification (Active Comparator): Individuals assigned to Arm 2 will undergo methadone detoxification as is standard procedure at the Rhode Island Department of Corrections. They will receive active assistance with returning to their home methadone clinic upon release from incarceration and 10 weeks financial assistance to pay for treatment.
  Interventions: Behavioral: Linkage to methadone maintenance

INTERVENTIONS:
Behavioral: Methadone Maintenance — Individuals who are enrolled in methadone maintenance treatment at the time of incarceration are maintained on pre-incarceration dosage levels of methadone during short-term (6 months or less)incarceration. They will be actively assisted to return to their home clinic upon release and receive 10 financial assistance with treatment payments.
  Arms: Methadone Maintenance
Behavioral: Linkage to methadone maintenance — Individuals in the comparison arm will undergo methadone detoxification during short term incarceration, however, they will be actively assisted to return to their home clinic upon release and receive 10 financial assistance with treatment payments.
  Arms: Methadone Detoxification

SUMMARY:
Methadone maintenance treatment (MMT) has been shown to be effective in reducing drug use, criminal activity and recidivism. Given this effectiveness, maintaining individuals who are enrolled in community MMT when committed to the Department of Corrections for short term incarceration would improve post release outcomes. However, this is rarely practiced in the United States. Current practice at the Rhode Island Department of Corrections is to detox inmates on methadone within 30 days of being incarcerated. More than 75% of these individuals are incarcerated for less than six months. The period immediately after release from incarceration is a particularly high-risk time for HIV and other problems including drug relapse and overdose.

The investigators hypothesize that inmates who are incarcerated for 6 months or less will have better outcomes and cost the state less money if they are maintained on their methadone dose and relinked to their community clinic at release, than the current practice of detoxification.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of maintaining methadone treatment during short-term incarceration vs. methadone detoxification on continuing treatment post release, relapse, reducing HIV risk behaviors and reincarceration. Persons who inject opiates are at increased risk for HIV through both injection and sexual practices. A substantial proportion of opiate addicted persons are incarcerated and a majority of the nearly 8 million individuals released from a correctional setting each year have a history of addiction. The period immediately after release from incarceration is a particularly high-risk time for HIV and other problems including drug relapse and overdose. Methadone is the most widely used opiate replacement therapy in the United States. Despite its demonstrated benefit in decreasing drug use, criminal activity, and recidivism, some individuals on methadone treatment are reincarcerated each year. More than 75% of those individuals are incarcerated for less than six months. A program that maintains these individuals at a therapeutic dose increases the likelihood that they will successfully return to treatment upon release.

The following primary specific aims will drive this research:

1. To determine the effect of maintaining methadone treatment during short-term incarceration vs. methadone detoxification on the time-to-post-release methadone treatment re-entry and relapse.
2. To determine whether maintaining methadone treatment during short-term incarceration is more effective in reducing HIV risk behaviors (both injecting and sexual) than methadone detoxification upon community re-entry.
3. To determine whether maintaining methadone treatment during short-term incarceration is more effective in reducing reincarceration than methadone detoxification.
4. To determine the impact on cost of the first three specific aims.

Secondary aims will include determining the effect of methadone maintenance during short-term incarceration versus methadone detoxification on:

* retention in community based methadone treatment;
* the number of fatal and nonfatal overdoses; and
* criminal behavior

The targeted population will be 300 recently incarcerated inmates enrolled in community methadone treatment at the time of incarceration. Follow-up interviews will occur 1-month post release from incarceration and 6, and 12 months from baseline at an independent study site. Both groups will receive a risk behavior reduction counseling intervention and linkage to community methadone treatment upon release. If this project is able to demonstrate that maintaining inmates on methadone for short-term incarcerations is effective, then this can influence correctional policy to work more collaboratively with community substance use treatment providers and to minimize disruption of treatment.

ELIGIBILITY:
Inclusion Criteria:

* currently incarcerated at the RI Department of Corrections
* enrolled in a Rhode Island methadone treatment program at the time of incarceration
* currently maintained at the pre-incarceration methadone dosage level
* estimated total incarceration time of < 6 months and > 1 week
* willing to be randomized and to conduct follow-up interviews for 12 months
* English or Spanish-speaking
* able to give informed consent
* age 18 years or older
* willing to remain on MMT and continue MMT after release.

Exclusion Criteria:

* pregnancy (pregnant women are maintained on pre-incarceration levels of methadone throughout their pregnancy for their health and the health of the fetus by the RI DOC, so are NOT eligible to be randomized to Arm 2)
* not fulfilling all of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Time to post release treatment engagement | 30 days post release
  Do individuals maintained on MMT during short term incarceration return to their community methadone clinic more rapidly than those who undergo methadone detoxification during short term incarceration? Individuals must return within 30 days of post release to be or be counted as not returning.
Reduction of HIV risk behaviors | 12 months
  To determine whether individuals maintained on MMT during short term incarceration report fewer HIV risk behaviors (both drug use and sexual) as compared to standard of care arm.
Time to relapse | 30 days post release
  To determine whether individuals maintained on MMT during short term incarceration report longer to relapse (or no relapse) to opiate use as compared to standard of care arm.
Cost effectiveness | 12 months
  To determine the costs, cost-effectiveness and cost-benefit associated with continuing methadone maintenance versus detoxification for jailed individuals. Variables to be assessed are: reincarceration, health care utilization (i.e. emergency room use, medications), subsidized housing,

SECONDARY OUTCOMES:
Treatment retention | 12 months
  length of time engaged in community methadone treatment
Fatal and nonfatal overdose | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Department of Corrections, Cranston, Rhode Island, United States

REFERENCES:
- [Derived] Rich JD, McKenzie M, Larney S, Wong JB, Tran L, Clarke J, Noska A, Reddy M, Zaller N. Methadone continuation versus forced withdrawal on incarceration in a combined US prison and jail: a randomised, open-label trial. Lancet. 2015 Jul 25;386(9991):350-9. doi: 10.1016/S0140-6736(14)62338-2. Epub 2015 May 28. PMID 26028120